CLINICAL TRIAL: NCT04112238
Title: Circulating Cell-free Tumor DNA and Metabolites in Cerebrospinal Fluid as Early Biomarkers of Secondary CNS Involvement in Diffuse Large B-cell Lymphoma
Brief Title: ctDNA and Metabolites in CSF as Early Biomarkers of Secondary CNS Involvement in Diffuse Large B-cell Lymphoma
Acronym: CNSctDNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Lars Møller Pedersen, Senior consultant, Herlev Hospital
Other Study IDs: CNSctDNA
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Diffuse Large B Cell Lymphoma; Central Nervous System Metastasis
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a prospective clinical study which investigates the use of new diagnostic methods to localize aggressive lymphoma involving the central nervous system(CNS). By measuring cell-free tumor DNA and metabolomics in cerebrospinal fluid and blood in patients with systemic Diffuse Large B-cell Lymphoma the investigators aim to improve the diagnostic certainty of an impending relapse of lymphoma in CNS.

DETAILED DESCRIPTION:
Diffuse Large B-cell Lymphoma is a malignant, aggressive cancer representing 40% of Non-Hodgkin Lymphomas globally. The risk of relapse after primary treatment is approximately 30% of which up to 10 % occurs in the central nervous system (CNS). The prognosis after CNS relapse is severely discouraging with an overall survival of 3-6 months. Currently CNS relapse is diagnosed by either flow cytometry performed on cerebrospinal fluid or a stereotactic biopsy based on tumor localization by an MRI scan. Both diagnostic methods however require a certain tumor mass in order avoid false negative test results.

The purpose of this study is to learn whether tumor-derived cell-free circulating DNA (cfDNA) and/or metabolite profiles from diffuse large B-cell lymphoma (DLBCL) cells can be identified in the cerebrospinal fluid (CSF), before the malignant cells themselves are detectable in CSF. Thus the investigators aim to investigate the diagnostic potential of cfDNA and/or metabolites measured in blood and cerebrospinal fluid. The study is based on the following four hypotheses:

Hypothesis 1: Measurement of cfDNA and/or metabolites in CSF are more sensitive methods of detecting DLBCL involvement in CNS compared to conventional diagnostics.

Hypothesis 2: Quantitative cfDNA/metabolomics in CSF has independent prognostic value in DLBCL.

Hypothesis 3: cfDNA and/or metabolite profile in CSF detected at primary diagnosis predicts relapse of DLBCL in the CNS also when CNS-IPI is taken into account.

Hypothesis 4: Particular aberrations of cfDNA and/or metabolite profiles detected in blood (plasma) may, in some cases, be associated with CNS involvement in DLBCL patients and/or predict CNS relapse.

The study is composed of a pilot study including 5 patients with verified either primary or secondary CNS lymphoma followed by two studies: One including 40 patients with de novo DLBCL and one including 30 patients in a relapse setting. The patients will have to consent to having a lumbar puncture performed and blood samples taken before treatment initiation. After treatment a second set of lumbar puncture and blood samples will be requested.

ELIGIBILITY:
Pilot Study:

Inclusion criteria:

1. Verified or suspected primary CNS lymphoma or verified or suspected DLBCL relapsed in the CNS
2. Treatment of the relapse not initiated (except pretreatment with corticosteroids)
3. Age ≥ 18 years
4. Patient must consent to genetic and metabolomic analysis of their cancer
5. Written informed consent

Exclusion criteria:

1. Evidence of a CNS mass creating mass-effect or midline shift such that lumbar puncture is contraindicated
2. Other contraindications to lumbar puncture according to local guidelines
3. Other previous or current hematological malignancy
4. Prior treatment for CNS disease (except CNS prophylaxis in first line lymphoma treatment)
5. Known CNS autoimmune or inflammatory disease
6. Known HIV infection
7. Patient is currently receiving treatment for DLBCL

Study 1

Inclusion criteria:

1. Previously diagnosed histologically documented DLBCL
2. Verified relapsed DLBCL
3. ≥ 1 prior DLBCL treatments
4. Treatment of the relapse not initiated (except pretreatment with corticosteroids)
5. Being able to undergo standard assessment ( eg, Fluorine-18 fluorodeoxyglucose positron emission tomography (18F-FDG-PET), MRI of the neuroaxis and bone marrow biopsy)
6. Tumor biopsy and/or bone-marrow biopsy used for diagnosis available
7. Age ≥ 18 years
8. ECOG performance status of 0, 1 or 2
9. Life expectancy ≥ 12 weeks
10. Patient must consent to permit genetic and metabolomic analysis of their cancer
11. Patient must consent to permit access to records in order to ascertain progression or relapse of their cancer
12. Written informed consent

Exclusion criteria:

1. Evidence of a CNS mass creating mass-effect or midline shift such that lumbar puncture is contraindicated
2. Other contraindications to lumbar puncture according to local guidelines
3. Other previous or current hematological malignancy
4. Previous or current primary CNS malignancy including know DLBCL relapse to the CNS
5. Prior treatment for CNS disease (except CNS prophylaxis in first line lymphoma treatment)
6. Known CNS autoimmune or inflammatory disease
7. Known HIV infection
8. Patient is currently receiving treatment for DLBCL (except pretreatment with corticosteroids)

Study 2

Inclusion criteria:

1. A newly diagnosed and histologically verified DLBCL
2. No prior DLBCL treatments
3. Anti-lymphoma treatment not initiated (except pretreatment with corticosteroids)
4. CNS-IPI >/= 3
5. Being able to undergo standard assessment ( eg, Fluorine-18 fluorodeoxyglucose positron emission tomography (18F-FDG-PET), MRI of the neuroaxis and bone marrow biopsy)
6. Tumor biopsy and/or bone-marrow biopsy used for diagnosis available
7. Age ≥ 18 years
8. ECOG performance status of 0, 1 or 2
9. Life expectancy >/= 12 weeks
10. Patient must consent to permit genetic analysis of their cancer
11. Patient must consent to permit access to records in order to ascertain progression or relapse of their cancer
12. Written informed consent

Exclusion criteria:

1. Evidence of a CNS mass creating mass-effect or midline shift such that lumbar puncture is contraindicated
2. Other contraindications to lumbar puncture according to local guidelines
3. Other previous or current hematological malignancy
4. Previous or current primary CNS malignancy including primary CNS lymphoma
5. Prior treatment for CNS disease
6. Known CNS autoimmune or inflammatory disease
7. Known HIV infection
8. Patient is currently receiving treatment for DLBCL (except pretreatment with corticosteroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See above
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-08-29 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
CSF tumor cfDNA and metabolite detectability and cytological/flow cytometric confirmation of CNS lymphoma at the time of diagnosis and relapse | Two years

SECONDARY OUTCOMES:
Progression free survival, PFS (time between inclusion and progression or relapse or beginning of a new treatment) | Two years
Overall survival, OS (time between inclusion and death) | Two years
Comparison of tumor cfDNA and metabolite levels and composition in CSF with levels in plasma at the time of diagnosis and relapse | Two years
For patients with both a pre- and a post-treatment CSF sample: correlation of cfDNA/metabolite levels pre-treatment to post-treatment with OS and risk of relapse. | Two years
Correlation of tumor cfDNA and metabolite levels and composition in CSF and patient survival at the time of diagnosis and relapse | Two years
Correlation of tumor cfDNA and/or metabolite identification in CSF of patients prior to diagnosis of CNS lymphoma at the time of diagnosis and relapse versus the appearance of later CNS lymphoma involvement | Two years
Comparison of the clonal similarity between tumor DNA in the blood and the CSF at relapse versus tumor DNA in the primary tumor (by NGS panel sequencing) | Two years
Comparison of CSF cytokines, other biomarkers and tumor DNA and metabolic profile in the prediction of CNS lymphoma disease | Two years
Comparison of mutational profile in diagnostic biopsy and/or cfDNA in peripheral blood with cfDNA in CSF and comparison of metabolic profiles in blood versus CSF in patients with and without development of CNS relapse. | Two years
YKL-40 in CSF as biomarker of CNS lymphoma | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Anne Elisabeth Reuben Tolley, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hopital, Herlev, Capital Region, Denmark